CLINICAL TRIAL: NCT02397915
Title: A Patient Preference Evaluation Study of Fluticasone Furoate Nasal Spray and Mometasone Furoate Nasal Spray in Subjects With Allergic Rhinitis
Brief Title: Patient Preference Study of Fluticasone Furoate and Mometasone Furoate Nasal Sprays
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 201474
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Rhinitis, Allergic, Perennial and Seasonal
Keywords: Nasal Spray; Fluticasone Furoate; Attributes; Single Dose; Allergic Rhinitis; Mometasone Furoate; Questionnaire; Preference
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone Furoate (Experimental): Subjects will receive a single dose of intranasal FF (total dose of 110 mcg) as 2 sprays per nostril / 4 sprays in total.
  Interventions: Drug: FF nasal spray
- Mometasone Furoate (Experimental): Subjects will receive a single dose of intranasal MF (total dose of 200 mcg) nasal spray as 2 sprays per nostril / 4 sprays in total.
  Interventions: Drug: MF nasal spray

INTERVENTIONS:
Drug: FF nasal spray — FF as a suspension for intranasal inhalation with unit dose strength of 27.5 mcg per dose x 4 doses (total dose 110 mcg) administered via a metered side-actuated nasal spray device.
  Arms: Fluticasone Furoate
Drug: MF nasal spray — MF as a suspension for intranasal inhalation with unit dose strength of 50 mcg per dose x 4 doses (total dose 200 mcg) administered via a metered top-actuated nasal spray device.
  Arms: Mometasone Furoate

SUMMARY:
The purpose of this study is to provide information on whether subjects with allergic rhinitis (AR) prefer the administration of fluticasone furoate (FF) nasal spray or mometasone furoate (MF) nasal spray based on how the products feel to the subjects when administered.

This Phase IV interventional study is a multi-center, randomized, double-blind, single-dose, cross-over subject preference study to evaluate and compare patient preference for FF [(total dose of 110 microgram (mcg)] and MF (total dose of 200 mcg) nasal sprays in subjects with allergic rhinitis. These two commonly used nasal sprays use different actuation systems (FF nasal spray is side-actuated; MF nasal spray is top-actuated) and this study will evaluate whether this difference is reflected in the patient-assessed attributes of the two nasal sprays. The attributes or properties which are being assessed by the subjects for these nasal sprays include smell, taste & aftertaste, drip down the throat, run out of the nose, urge to sneeze, and irritation.

The single-day study per subject comprises screening and all treatments and procedures. Eligible subjects will be randomized 1:1 to a cross-over treatment schedule so that all subjects receive both products. One group of subjects will have two sprays of FF administered in each nostril whilst a second group will have two sprays of MF administered into each nostril. At 30 (± 5) minutes after the first study medication treatment, the two groups will switch. The first group will then have two sprays of MF administered into each nostril and the second group will then have two sprays of FF administered into each nostril. After each treatment the subject will complete two sets of attributes questionnaires ('immediate' and 'delayed'). A subject-rated 'immediate' attributes questionnaire will be completed immediately following each treatment and a subject-rated 'delayed' attributes questionnaire will be completed approximately 2 minutes after each treatment. Upon completion of the second set of these two attributes questionnaires (immediate and delayed), a preference questionnaire will be completed by the subject. In the preference questionnaire, the subject states their preferred treatment, if any, for each of the product attributes, and finally states their overall preferred treatment, if any.

There will be follow-up contact with the subject 24 (± 4) and 96 (± 4) hours after administration of the last treatment. The study is planned to enroll about 300 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are between 18 to 65 years of age, inclusive at the time of signing the informed consent.
* Severity of disease: Subjects who meet the below criteria and who may also have vasomotor rhinitis are eligible for the study. A positive skin test to perennial (for example, but not limited to, animal dander, house dust mites, cockroach, mould) and / or seasonal (for example, but not limited to, grass, tree, weed, ragweed) allergen within 12 months prior to Screening. If a subject has not been tested in the 12 months prior to Screening, a positive skin test (by prick method) is required at Screening. A positive skin test is defined as a wheal >=3 millimeters (mm) larger than the diluent control for prick testing. In vitro tests for specific Immunoglobulin E (IgE) [such as radioallergosorbent test (RAST), paper radioimmunosorbent test (PRIST)] will not be allowed as a diagnosis of AR.
* A female subject is eligible to participate if she is not pregnant [as confirmed by a negative urine (preferred) or serum human chorionic gonadotrophin (hCG) test], not lactating, and at least one of the following conditions applies: (a) Non-reproductive potential defined as premenopausal females with a documented tubal ligation or documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion or hysterectomy or documented bilateral oophorectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. (b) Reproductive potential and agrees to follow one of the options listed below in the GlaxoSmithKline (GSK) modified list of highly effective methods for avoiding pregnancy in females of reproductive potential (FRP) requirements from 30 days prior to the first dose of study medication and until at least 4 days after the last dose of study medication. The GSK modified list of highly effective methods includes: contraceptive subdermal implant that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Oral contraceptive; either combined or progestogen alone; Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches; Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject. This list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis.
* A male subject is eligible to participate if (a) subjects with female partners of child bearing potential comply with the following contraception requirements from the time of first dose of study medication until at least 4 days after the last dose of study medication; (b) Vasectomy with documentation of azoospermia; (c) Male condom plus partner use of one of the contraceptive options: Contraceptive subdermal implant that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Oral contraceptive, either combined or progestogen alone, Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches. These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Understanding of questionnaires: In the opinion of the investigator, subject possesses a degree of understanding of the written questionnaires that enables the subject to complete study participation.
* Informed consent: Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

* Concurrent conditions / Medical History: Concomitant medical conditions defined as but not limited to a historical or current evidence of clinically significant uncontrolled disease of any body system (e.g., tuberculosis, psychological disorders, eczema, uncontrolled diabetes, immunosuppression). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through study participation, or compromise the scientific validity of the study; A respiratory infection at time of study participation; A condition associated with anosmia (loss of smell) and ageusia (loss of taste) within 2 weeks of study - may be self-reported condition experienced by the subject; Clinical evidence of a Candida infection of the nose or oropharynx; Acute rhinosinusitis within 60 days of screening; Current severe physical obstruction of the nose (e.g., deviated septum or nasal polyp) or nasal septal perforation or nasal trauma or nasal ulcers; History of haemorrhagic diathesis, atrophic rhinitis, or recurrent nasal bleeding which may, in the opinion of the investigator, impact on the safety of the subject or the scientific validity of the study; Nasal biopsy within 60 days of screening; Nasal jewellery or piercings which could impact nasal safety or airway resistance; Rhinitis medicamentosa within 60 days of screening; History of glaucoma, cataracts or raised intraocular pressure.
* Concomitant medications: Use of intranasal corticosteroids (FF, MF or others) within 4 weeks of study participation; Recent or ongoing use of a corticosteroid by a non-nasal route which, in the opinion of the investigator, could preclude subject participation in the study; Use of intranasal medications (including intranasal antihistamines, intranasal decongestants, intranasal saline) within 1 week of study participation; Use of medications which, in the opinion of the investigator, could disturb the taste or smell faculties of the subject; Use of any medications that significantly inhibit the cytochrome P450 (CYP) sub-family CYP3A4, including but not limited to ritonavir and ketoconazole, within 4 weeks of study participation.
* Relevant habits: Use of perfume or strong-smelling cosmetic products or oral rinse or similar products on the study day that could, in the opinion of the investigator, compromise participation in the study. Subjects should be notified of this criterion prior to study participation; Use of tobacco, or inhaled or oral nicotine-containing products, is not allowed for 12 hours prior to the start of dosing.
* Contraindications: History of sensitivity to any of the study procedures or medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Diagnostic assessments and other criteria: Positive pregnancy test or female who is breastfeeding; The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer), unless more stringent local guidelines need to be followed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2015-06-08 (Actual); Study Completion 2015-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Argentina (2):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
- Australia (3):
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, Maroubra, New South Wales
  - GSK Investigational Site, Murdoch, Western Australia
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Stavropol
- South Korea (3):
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seongnam-si, Gyeonggi-do
  - GSK Investigational Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Meltzer EO, Bardelas J, Goldsobel A, Kaiser H. A preference evaluation study comparing the sensory attributes of mometasone furoate and fluticasone propionate nasal sprays by patients with allergic rhinitis. Treat Respir Med. 2005;4(4):289-96. doi: 10.2165/00151829-200504040-00007. PMID 16086602
- [Background] Meltzer EO, Stahlman JE, Leflein J, Meltzer S, Lim J, Dalal AA, Prillaman BA, Philpot EE. Preferences of adult patients with allergic rhinitis for the sensory attributes of fluticasone furoate versus fluticasone propionate nasal sprays: a randomized, multicenter, double-blind, single-dose, crossover study. Clin Ther. 2008 Feb;30(2):271-9. doi: 10.1016/j.clinthera.2008.02.005. PMID 18343265
- [Background] Sher ER, Ross JA. Intranasal corticosteroids: the role of patient preference and satisfaction. Allergy Asthma Proc. 2014 Jan-Feb;35(1):24-33. doi: 10.2500/aap.2014.35.3725. PMID 24433594
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 201474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-dose, cross-over participant (par.) preference study, where participants with seasonal allergic rhinitis or perennial allergic rhinitis were randomized, in ratio of 1:1, to receive fluticasone furoate (FF) nasal spray and mometasone furoate (MF) nasal spray.
Groups:
- Period 1: FF 110 µg: Participants received two sprays of FF (total dose of 110 micrograms [µg]) in each nostril (total 4 sprays). Two study treatments were administered 30 minutes (+/- 5) apart by a third party administrator using a metered nasal spray.
- Period 1: MF 200 µg: Participants received two sprays of MF (total dose of 200 µg) in each notstril (total 4 sprays). Two study treatments were administered 30 minutes (+/- 5) apart by a third party administrator using a metered nasal spray.
- Period 2: MF 200 µg: Participants received two sprays of MF (total dose of 200 µg) in each nostril (total 4 sprays).
- Period 2: FF 110 µg: Participants received FF (total dose of 110 µg) in each nostril (total 4 sprays).
Period: Period 1
Arm/Group | Period 1: FF 110 µg | Period 1: MF 200 µg | Period 2: MF 200 µg | Period 2: FF 110 µg
Started | 150 | 150 | 0 | 0
Completed | 149 | 149 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Period 1: FF 110 µg | Period 1: MF 200 µg | Period 2: MF 200 µg | Period 2: FF 110 µg
Started | 0 | 0 | 149 | 149
Completed | 0 | 0 | 149 | 149
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FF 110 µg /MF 200 µg or MF 200 µg /FF 110 µg: All participants received treatments in one of two treatment sequences, Sequence 1: two sprays of FF (total of 110 µg) in each nostril (total 4 sprays) in Period 1 and two sprays of MF (total of 200 µg) in each nostril (total 4 sprays) in Period 2; Sequence 2: FF (110 µg) followed by MF (total of 200 µg) and MF (total of 200 µg) followed by FF (110 µg) in Period 2. Two study treatments were administered 30 minutes (+/-5) apart by a third party administrator using a metered nasal spray.
Arm/Group | FF 110 µg /MF 200 µg or MF 200 µg /FF 110 µg
Number analyzed (Participants) | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.4 (13.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185
  Male | 115
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian Heritage | 49
  Asian - South East Asian Heritage | 19
  Asian - Mixed Race | 7
  Native Hawaiian or other Pacific Islander | 2
  White - Arabic/North African Heritage | 2
  White - White/Caucasian/European Heritage | 217
  Mixed Race | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Preference for Nasal Spray Assessed by Preference Questionnaire.
Description: An overall preference questionnaire (OPQ) was used to evaluate participants' preference for nasal spray therapy for the given treatments. OPQ allows the responder three options, based on products attributes, i.e. preference for product 1; preference for product 2 and no preference. The OPQ was completed by each participant approximately 4 minutes after administration of the second treatment in Period 2. Overall participant preferences were analyzed using Prescott's test, as approximated by a Cochran-Mantel-Haenszel (CMH) test, adjusted for country and symptomatology. All preference p-values were also adjusted for multiplicity using Hochberg's method.
Time Frame: Approximately four minutes after the administration of the second treatment
Population: Per Protocol (PP) Population: comprised of all participants who completed both treatment Periods and the questionnaires associated with them.
Measure: Number; unit: Participants
Groups:
- FF 110 µg /MF 200 µg: Participants received two sprays of FF (total dose of 110 µg) in each nostril (total 4 sprays) in Period 1 followed by two sprays of MF (total dose of 200 µg) in each nostril (total 4 sprays) in Period 2. Two study treatments were administered 30 minutes (+/- 5) apart by a third party administrator using a metered nasal spray.
- MF 200 µg /FF 110 µg: Participants received two sprays of MF (total dose of 200 µg) in each notstril (total 4 sprays) in Period 1 followed by two sprays of FF (total dose of 110 µg) in each nostril (total 4 sprays) in Period 2. Two study treatments were administered 30 minutes (+/- 5) apart by a third party administrator using a metered nasal spray.
Arm/Group | FF 110 µg /MF 200 µg | MF 200 µg /FF 110 µg
Number analyzed (Participants) | 138 | 138
Participants
  FF 110 µg | 96 | 59
  MF 200 µg | 30 | 57
  No preference | 12 | 22
Statistical Analysis 1: Comparison: FF 110 µg /MF 200 µg vs MF 200 µg /FF 110 µg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Par. preferences were analyzed using Prescott's test, as approximated by a Cochran-Mantel-Haenszel test, adjusted for country and symptomatology. All preference p-values were also adjusted for multiplicity using Hochberg's method

2. Secondary Outcome: Number of Participants With Preference for Individual Nasal Spray Attributes Assessed by Preference Questionnaire
Description: An overall preference questionnaire (OPQ) was used to evaluate participants' attribute preference for nasal spray therapy for the given treatment. OPQ allows the responder three options, based on products attributes, i.e. preference for product 1; preference for product 2 and no preference. Products attributes included scent/odor, immediate taste, after taste, less drip through throat (LDTT), less run out of nose (LRON), more soothing, less irritating and urge to sneeze (UTS). The OPQ was completed by each participant approximately 4 minutes after administration of the second treatment (tmt) in Period 2. Overall participant preferences were analyzed using Prescott's test, as approximated by a Cochran-Mantel-Haenszel (CMH) test, adjusted for country (ctry) and symptomatology (sym). All preference p-values were also adjusted for multiplicity using Hochberg's method.
Time Frame: Approximately four minutes after the administration of the second treatment
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg /MF 200 µg | MF 200 µg /FF 110 µg
Number analyzed (Participants) | 138 | 138
Participants
  Scent/odor, FF110 µg | 53 | 28
  Scent/odor, MF 200 µg | 21 | 31
  Scent/odor, no preference | 64 | 79
  Immediate taste, FF110 µg | 35 | 25
  Immediate taste, MF 200 µg | 22 | 27
  Immediate taste, no preference | 81 | 86
  After taste, FF110 µg | 41 | 28
  After taste, MF 200 µg | 21 | 28
  After taste, no preference | 76 | 82
  LDTT, FF110 µg | 65 | 37
  LDTT, MF 200 µg | 15 | 36
  LDTT, no preference | 58 | 65
  LRON, FF110 µg | 60 | 34
  LRON, MF 200 µg | 22 | 37
  LRON, no preference | 56 | 67
  More soothing, FF110 µg | 68 | 53
  More soothing, MF 200 µg | 35 | 47
  More soothing, no preference | 35 | 38
  Less irritating, FF110 µg | 68 | 37
  Less irritating, MF 200 µg | 12 | 33
  Less irritating, no preference | 58 | 68
  UTS, FF110 µg | 19 | 22
  UTS, MF 200 µg | 19 | 17
  UTS, no preference | 100 | 99
Statistical Analysis 1: Comparison: FF 110 µg /MF 200 µg vs MF 200 µg /FF 110 µg; Test type: Superiority or Other; p = 0.065, Cochran-Mantel-Haenszel — Par. preferences were analyzed using Prescott's test, as approximated by a CMH test, adjusted for ctry and sym. All preference p-values were also adjusted for multiplicity using Hochberg's method. P-value is for product attribute scent/odor
Statistical Analysis 2: Comparison: FF 110 µg /MF 200 µg vs MF 200 µg /FF 110 µg; Test type: Superiority or Other; p = 0.532, Cochran-Mantel-Haenszel — Par. preferences were analyzed using Prescott's test, as approximated by a CMH test, adjusted for ctry and sym. All preference p-values were also adjusted for multiplicity using Hochberg's method. P-value is for product attribute immediate taste
Statistical Analysis 3: Comparison: FF 110 µg /MF 200 µg vs MF 200 µg /FF 110 µg; Test type: Superiority or Other; p = 0.138, Cochran-Mantel-Haenszel — Par. preferences were analyzed using Prescott's test, as approximated by a CMH test, adjusted for ctry and sym. All preference p-values were also adjusted for multiplicity using Hochberg's method. P-value is for product attribute after taste
Statistical Analysis 4: Comparison: FF 110 µg /MF 200 µg vs MF 200 µg /FF 110 µg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Par. preferences were analyzed using Prescott's test, as approximated by a CMH test, adjusted for ctry and sym. All preference p-values were also adjusted for multiplicity using Hochberg's method. P-value is for product attribute LDTT
Statistical Analysis 5: Comparison: FF 110 µg /MF 200 µg vs MF 200 µg /FF 110 µg; Test type: Superiority or Other; p = 0.017, Cochran-Mantel-Haenszel — Par. preferences were analyzed using Prescott's test, as approximated by a CMH test, adjusted for ctry and sym. All preference p-values were also adjusted for multiplicity using Hochberg's method. P-value is for product attribute LRON
Statistical Analysis 6: Comparison: FF 110 µg /MF 200 µg vs MF 200 µg /FF 110 µg; Test type: Superiority or Other; p = 0.046, Cochran-Mantel-Haenszel — Par. preferences were analyzed using Prescott's test, as approximated by a CMH test, adjusted for ctry and sym. All preference p-values were also adjusted for multiplicity using Hochberg's method. P-value is for product attribute more soothing
Statistical Analysis 7: Comparison: FF 110 µg /MF 200 µg vs MF 200 µg /FF 110 µg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Par. preferences were analyzed using Prescott's test, as approximated by a CMH test, adjusted for ctry and sym. All preference p-values were also adjusted for multiplicity using Hochberg's method. P-value is for product attribute less irritating
Statistical Analysis 8: Comparison: FF 110 µg /MF 200 µg vs MF 200 µg /FF 110 µg; Test type: Superiority or Other; p = 0.532, Cochran-Mantel-Haenszel — Par. preferences were analyzed using Prescott's test, as approximated by a CMH test, adjusted for ctry and sym. All preference p-values were also adjusted for multiplicity using Hochberg's method. P-value is for product attribute UTS

3. Secondary Outcome: Number of Participants Responding to the Immediate Attributes Question Regarding Scent/Odor
Description: Immediate attributes questionnaire was used to evaluate immediate ratings of participant for individual attributes of FF and MF nasal spray. Number of participants responding to product attributes i.e. scent/odor, using immediate attributes questionnaire, Question 1, "Did product have a scent/odor?" are summarized. The immediate attributes questionnaire was completed immediately following each treatment in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: none; 1: very mild; 2: mild; 3: neither mild nor strong; 4: slightly strong; 5; moderately strong; 6: very strong. Immediate attribute ratings were analyzed using an analysis of variance (ANOVA) mixed model with participant as a random effect, and country, treatment, period, and Baseline (BL) rhinitis symptomatology subgroup (subgrp), and treatment sequence as main effects. P-values associated with tests of immediate attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Immediately following each treatment in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Groups:
- FF 110 µg: Participants received two sprays of FF (total dose of 110 µg) in each nostril (total 4 sprays) by the third party administrator using metered nasal spray.
- MF 200 µg: Participants received two sprays of MF (total of 200 µg) in each nostril (total 4 sprays) by the third party administrator using metered nasal spray.
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  None | 180 | 185
  Very mild | 60 | 59
  Mild | 24 | 16
  Neither mild nor strong | 2 | 2
  Slightly strong | 8 | 11
  Moderately strong | 2 | 3
  Very strong | 0 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel — Analyzed using an ANOVA mixed model with par. as random effect, ctry, tmt, BL rhinitis sym subgrp, and tmt seq as main effects. P-values for all immediate attribute rating scores adjusted for multiplicity using Hochberg's method; Median Difference (Final Values) = 0.00

4. Secondary Outcome: Number of Participants Responding to the Immediate Attributes Question Regarding Satisfaction With Scent/Odor
Description: Immediate attributes questionnaire (ques) was used to evaluate immediate ratings of par. for individual attributes of FF and MF nasal spray. Number of par. responding to product attributes i.e. scent/odor, using immediate attributes ques, Question 2, "How satisfied with scent/odor?" are summarized. The immediate' attributes ques was completed immediately following each treatment (trt) in Period 1 and 2. Par. specified their responses on a 6-point scale: 0: very satisfied; 1: moderately satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied; 5; moderately dissatisfied; 6: very dissatisfied. Immediate attribute ratings were analyzed using an analysis of variance mixed model with par. as a random effect, and country, trt, period, and BL rhinitis symptomatology subgroup, and trt sequence as main effects. P-values associated with tests of immediate attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Immediately following each treatment in Period 1 and 2
Population: PP Population. Only participants responded to the question were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 96 | 91
Participants
  Very satisfied | 29 | 24
  Moderately satisfied | 19 | 27
  Somewhat satisfied | 10 | 14
  Neither satisfied nor dissatisfied | 27 | 17
  Somewhat dissatisfied | 7 | 3
  Moderately dissatisfied | 2 | 4
  Very dissatisfied | 2 | 2
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 1.00, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Median Difference (Final Values) = 0.00

5. Secondary Outcome: Number of Participants Responding to the Immediate Attributes Question Regarding Satisfaction Not to Have Scent/Odor
Description: Immediate attributes questionnaire was used to evaluate immediate ratings of par. for individual attributes of FF and MF nasal spray. Number of par. responding to product attributes i.e. scent/odor, using immediate attributes questionnaire, Question 3, "How satisfied not to have scent/odor?" are summarized. The immediate' attributes questionnaire was completed immediately following each trt in Period 1 and 2. Par. specified their responses on a 6-point scale: 0: very satisfied; 1: moderately satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied; 5; moderately dissatisfied; 6: very dissatisfied. Immediate attribute ratings were analyzed using an analysis of variance mixed model with par. as a random effect, and country, trt, period, and BL rhinitis symptomatology subgroup, and trt sequence as main effects. P-values associated with tests of immediate attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Immediately following each treatment in Period 1 and 2
Population: PP Population. Only participants responded to the question were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 182 | 186
Participants
  Very satisfied | 135 | 132
  Moderately satisfied | 19 | 19
  Somewhat satisfied | 7 | 8
  Neither satisfied nor dissatisfied | 16 | 21
  Somewhat dissatisfied | 1 | 3
  Moderately dissatisfied | 3 | 2
  Very dissatisfied | 1 | 1
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 1.00, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Median Difference (Final Values) = 0.00

6. Secondary Outcome: Number of Participants Responding to the Immediate Attributes Question Regarding Immediate Taste.
Description: Immediate attributes questionnaire was used to evaluate immediate ratings of participant for individual attributes of FF and MF nasal spray. Number of participants responding to product attributes i.e. taste, using immediate attributes questionnaire, Question 4, "Did product have an immediate taste?" are summarized. The immediate attributes questionnaire was completed immediately following each treatment in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: no; 1: very mild; 2: mild; 3: neither mild nor strong; 4: slightly strong; 5; moderately strong; 6: very strong. Immediate attribute ratings were analyzed using an analysis of variance mixed model with participant as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of immediate attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Immediately following each treatment in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  No | 226 | 205
  Very mild | 34 | 40
  Mild | 9 | 20
  Neither mild nor strong | 0 | 0
  Slightly strong | 4 | 10
  Moderately strong | 3 | 0
  Very strong | 0 | 1
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 0.179, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Median Difference (Final Values) = 0.00

7. Secondary Outcome: Number of Participants Responding to the Immediate Attributes Question Regarding Satisfaction With Immediate Taste.
Description: Immediate attributes questionnaire was used to evaluate immediate ratings of par. for individual attributes of FF and MF nasal spray. Number of par. responding to product attributes i.e. taste, using immediate attributes questionnaire, Question 5, "How satisfied with immediate taste?" are summarized. The immediate attributes questionnaire was completed immediately following each treatment in Period 1 and 2. Par. specified their responses on a 6-point scale: 0: very satisfied; 1: moderately satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied; 5; moderately dissatisfied; 6: very dissatisfied. Immediate attribute ratings were analyzed using an analysis of variance mixed model with par. as a random effect, and country, treatment, period, and BL rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of immediate attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Immediately following each treatment in Period 1 and 2
Population: PP Population. Only participants responded to the question were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 50 | 71
Participants
  Very satisfied | 14 | 16
  Moderately satisfied | 14 | 11
  Somewhat satisfied | 5 | 10
  Neither satisfied nor dissatisfied | 10 | 22
  Somewhat dissatisfied | 3 | 5
  Category title 6. Moderately dissatisfied | 2 | 5
  Very dissatisfied | 2 | 2
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 1.00, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Median Difference (Final Values) = 0.00

8. Secondary Outcome: Number of Participants Responding to the Immediate Attributes Question Regarding Medicine Running Down Throat
Description: Immediate attributes questionnaire was used to evaluate immediate ratings of participant for individual attributes of FF and MF nasal spray. Number of participants responding to product attributes using immediate attributes questionnaire, Question 6, "Did medicine run down throat?" are summarized. The immediate attributes questionnaire was completed immediately following each treatment in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: none; 1: very slightly; 2: slightly; 3: neither slightly nor moderately; 4: moderately; 5; markedly; 6: very markedly. Immediate attribute ratings were analyzed using an analysis of variance mixed model with participant as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of immediate attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Immediately following each treatment in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  None | 197 | 158
  Very slightly | 56 | 64
  Slightly | 15 | 33
  Neither slightly nor moderately | 2 | 5
  Moderately | 4 | 10
  Markedly | 1 | 4
  Very markedly | 1 | 2
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Median Difference (Final Values) = 0.00

9. Secondary Outcome: Number of Participants Responding to the Immediate Attributes Question Regarding Medicine Running Out of Nose.
Description: Immediate attributes questionnaire was used to evaluate immediate ratings of participant for individual attributes of FF and MF nasal spray. Number of participants responding to product attributes using immediate attributes questionnaire, Question 7, "Did medicine run out of nose?" are summarized. The immediate attributes questionnaire was completed immediately following each treatment in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: none; 1: very slightly; 2: slightly; 3: neither slightly nor moderately; 4: moderately; 5; markedly; 6: very markedly. Immediate attribute ratings were analyzed using an analysis of variance mixed model with participant as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of immediate attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Immediately following each treatment in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  None | 169 | 147
  Very slightly | 80 | 75
  Slightly | 21 | 29
  Neither slightly nor moderately | 3 | 6
  Moderately | 3 | 12
  Markedly | 0 | 5
  Very markedly | 0 | 2
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Median Difference (Final Values) = 0.00

10. Secondary Outcome: Number of Participants Responding to the Immediate Attributes Question Regarding Soothing
Description: Immediate attributes questionnaire was used to evaluate immediate ratings of participant for individual attributes of FF and MF nasal spray. Number of participants responding to product attributes using immediate attributes questionnaire, Question 8, "Did product feel soothing?" are summarized. The immediate attributes questionnaire was completed immediately following each treatment in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: none; 1: very slightly; 2: slightly; 3: neither slightly nor moderately; 4: moderately; 5; markedly; 6: very markedly. Immediate attribute ratings were analyzed using an analysis of variance mixed model with participant as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of immediate attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Immediately following each treatment in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  None | 59 | 67
  Very slightly | 62 | 65
  Slightly | 49 | 41
  Neither slightly nor moderately | 30 | 28
  Moderately | 34 | 41
  Markedly | 29 | 23
  Very markedly | 13 | 11
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Median Difference (Final Values) = 0.00

11. Secondary Outcome: Number of Participants Responding to the Immediate Attributes Question Regarding Sneezing
Description: Immediate attributes questionnaire was used to evaluate immediate ratings of par. for individual attributes of FF and MF nasal spray. Number of par. responding to product attributes using immediate attributes questionnaire, Question 9, "Did product make want to sneeze?" are summarized. The immediate attributes questionnaire was completed immediately following each treatment in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: no urgency; 1: very slightly urgency; 2: slightly urgency; 3: neither slightly nor moderately urgency; 4: moderately urgency; 5; markedly urgency; 6: very markedly urgency. Immediate attribute ratings were analyzed using an analysis of variance mixed model with par. as a random effect, and country, treatment, period, and BL rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of immediate attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Immediately following each treatment in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  No urgency | 249 | 233
  Very slightly urgency | 13 | 21
  Slightly urgency | 8 | 12
  Neither slightly nor moderately urgency | 1 | 1
  Moderately urgency | 5 | 6
  Markedly urgency | 0 | 2
  Very markedly urgency | 0 | 1
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 0.188, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Median Difference (Final Values) = 0.00

12. Secondary Outcome: Number of Participants Responding to the Delayed Attributes Question Regarding Scent/Odor.
Description: Delayed attributes questionnaire was used to evaluate immediate ratings of participant for individual attributes of FF and MF nasal spray. Number of participants responding to product attributes i.e. scent/odor, using delayed attributes questionnaire, Question 1, "Did product have a scent/odor?" are summarized. The delayed attributes questionnaire was completed 2 minutes after dosing, in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: none; 1: very mild; 2: mild; 3: neither mild nor strong; 4: slightly strong; 5; moderately strong; 6: very strong. Delayed attribute ratings were analyzed using an analysis of variance mixed model with participant as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of delayed attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Approximatly two minutes after the dosing in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  None | 209 | 220
  Very mild | 48 | 36
  Mild | 15 | 12
  Neither mild nor strong | 0 | 4
  Slightly strong | 3 | 3
  Moderately strong | 1 | 1
  Very strong | 0 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 0.951, Cochran-Mantel-Haenszel — Analyzed using an ANOVA mixed model with par. as random effect, ctry, tmt, BL rhinitis sym subgrp, and tmt seq as main effects. P-values for all delayed attribute rating scores adjusted for multiplicity using Hochberg's method; Median Difference (Final Values) = 0.00

13. Secondary Outcome: Number of Participants Responding to the Delayed Attributes Question Regarding Satisfaction With Scent/Odor.
Description: Delayed attributes questionnaire was used to evaluate delayed ratings of par. for individual attributes of FF and MF nasal spray. Number of par. responding to product attributes i.e. scent/odor, using delayed attributes questionnaire, Question 2, "How satisfied with scent/odor?" are summarized. The delayed attributes questionnaire was completed 2 minutes after dosing, in Period 1 and 2. Par. specified their responses on a 6-point scale: 0: very satisfied; 1: moderately satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied; 5; moderately dissatisfied; 6: very dissatisfied. Delayed attribute ratings were analyzed using an analysis of variance mixed model with par. as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of delayed attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Approximatly two minutes after the dosing in Period 1 and 2
Population: PP Population. Only participants responded to the question were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 67 | 56
Participants
  Very satisfied | 19 | 13
  Moderately satisfied | 18 | 16
  Somewhat satisfied | 9 | 7
  Neither satisfied nor dissatisfied | 15 | 14
  Somewhat dissatisfied | 3 | 4
  Moderately dissatisfied | 1 | 2
  Very dissatisfied | 2 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 0.951, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Median Difference (Final Values) = 0.00

14. Secondary Outcome: Number of Participants Responding to the Delayed Attributes Question Regarding Satisfaction Not to Have Scent/Odor.
Description: Delayed attributes questionnaire was used to evaluate delayed ratings of par. for individual attributes of FF and MF nasal spray. Number of par. responding to product attributes i.e. scent/odor, using delayed attributes questionnaire, Question 3, "How satisfied not to have scent/odor?" are summarized. The delayed attributes questionnaire was completed 2 minutes after dosing, in Period 1 and 2. Par. specified their responses on a 6-point scale: 0: very satisfied; 1: moderately satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied; 5; moderately dissatisfied; 6: very dissatisfied. Delayed attribute ratings were analyzed using an analysis of variance mixed model with par. as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of delayed attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Approximatly two minutes after the dosing in Period 1 and 2
Population: PP Population. Only participants responded to the question were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 210 | 221
Participants
  Very satisfied | 150 | 151
  Moderately satisfied | 25 | 28
  Somewhat satisfied | 11 | 12
  Neither satisfied nor dissatisfied | 19 | 25
  Somewhat dissatisfied | 1 | 2
  Moderately dissatisfied | 2 | 1
  Very dissatisfied | 2 | 2
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 0.951, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Median Difference (Final Values) = 0.00

15. Secondary Outcome: Number of Participants Responding to the Delayed Attributes Question Regarding Aftertaste.
Description: Delayed attributes questionnaire was used to evaluate delayed ratings of participant for individual attributes of FF and MF nasal spray. Number of participants responding to product attributes i.e. taste, using delayed attributes questionnaire, Question 4, "Did product have an aftertaste?" are summarized. The delayed attributes questionnaire was completed 2 minutes after dosing, in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: no; 1: very mild; 2: mild; 3: neither mild nor strong; 4: slightly strong; 5; moderately strong; 6: very strong. Immediate attribute ratings were analyzed using an analysis of variance mixed model with participant as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of delayed attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Approximatly two minutes after the dosing in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  No | 217 | 185
  Very mild | 42 | 61
  Mild | 13 | 17
  Neither mild nor strong | 2 | 4
  Slightly strong | 1 | 7
  Moderately strong | 1 | 2
  Very strong | 0 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Median Difference (Final Values) = 0.00

16. Secondary Outcome: Number of Participants Responding to the Delayed Attributes Question Regarding Satisfaction With Aftertaste.
Description: Delayed attributes questionnaire was used to evaluate delayed ratings of par. for individual attributes of FF and MF nasal spray. Number of par. responding to product attributes i.e. taste, using delayed attributes questionnaire, Question 5, "How satisfied with aftertaste?" are summarized. The delayed attributes questionnaire was completed 2 minutes after dosing, in Period 1 and 2. Par. specified their responses on a 6-point scale: 0: very satisfied; 1: moderately satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied; 5; moderately dissatisfied; 6: very dissatisfied. Delayed attribute ratings were analyzed using an analysis of variance mixed model with par. as a random effect, and country, treatment, period, and BL rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of delayed attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Approximatly two minutes after the dosing in Period 1 and 2
Population: PP Population. Only participants responded to the question were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 62 | 92
Participants
  Very satisfied | 20 | 18
  Moderately satisfied | 13 | 22
  Somewhat satisfied | 11 | 12
  Neither satisfied nor dissatisfied | 13 | 25
  Somewhat dissatisfied | 2 | 10
  Moderately dissatisfied | 3 | 4
  Very dissatisfied | 0 | 1
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 0.223, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Median Difference (Final Values) = 0.00

17. Secondary Outcome: Number of Participants Responding to the Delayed Attributes Question Regarding Medicine Running Down Throat.
Description: Delayed attributes questionnaire was used to evaluate delayed ratings of participant for individual attributes of FF and MF nasal spray. Number of participants responding to product attributes using delayed attributes questionnaire, Question 6, "Did medicine run down throat?" are summarized. The delayed attributes questionnaire was completed 2 minutes after dosing, in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: none; 1: very slightly; 2: slightly; 3: neither slightly nor moderately; 4: moderately; 5; markedly; 6: very markedly. Delayed attribute ratings were analyzed using an analysis of variance mixed model with participant as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of delayed attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Approximatly two minutes after the dosing in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  None | 188 | 147
  Very slightly | 57 | 73
  Slightly | 24 | 33
  Neither slightly nor moderately | 2 | 5
  Moderately | 3 | 12
  Markedly | 2 | 5
  Very markedly | 0 | 1
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Median Difference (Final Values) = 0.00

18. Secondary Outcome: Number of Participants Responding to the Delayed Attributes Question Regarding Smedicine Running Out of Nose.
Description: Delayed attributes questionnaire was used to evaluate delayed ratings of participant for individual attributes of FF and MF nasal spray. Number of participants responding to product attributes using delayed attributes questionnaire, Question 7, "Did medicine run out of nose?" are summarized. The delayed attributes questionnaire was completed 2 minutes after dosing, in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: none; 1: very slightly; 2: slightly; 3: neither slightly nor moderately; 4: moderately; 5; markedly; 6: very markedly. Delayed attribute ratings were analyzed using an analysis of variance mixed model with participant as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of delayed attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Approximatly two minutes after the dosing in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  None | 186 | 165
  Very slightly | 68 | 69
  Slightly | 16 | 30
  Neither slightly nor moderately | 2 | 4
  Moderately | 4 | 7
  Markedly | 0 | 1
  Very markedly | 0 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 0.008, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Median Difference (Final Values) = 0.00

19. Secondary Outcome: Number of Participants Responding to the Delayed Attributes Question Regarding Soothing.
Description: Delayed attributes questionnaire was used to evaluate delayed ratings of participant for individual attributes of FF and MF nasal spray. Number of participants responding to product attributes using delayed attributes questionnaire, Question 8, "Did product feel soothing?" are summarized. The delayed attributes questionnaire was completed 2 minutes after dosing, in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: none; 1: very slightly; 2: slightly; 3: neither slightly nor moderately; 4: moderately; 5; markedly; 6: very markedly. Delayed attribute ratings were analyzed using an analysis of variance mixed model with participant as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of delayed attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Approximatly two minutes after the dosing in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  None | 65 | 62
  Very slightly | 53 | 65
  Slightly | 48 | 47
  Neither slightly nor moderately | 29 | 28
  Moderately | 38 | 46
  Markedly | 29 | 19
  Very markedly | 14 | 9
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 0.831, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Median Difference (Final Values) = 0.00

20. Secondary Outcome: Number of Participants Responding to the Delayed Attributes Question Regarding Nasal Irritation.
Description: Delayed attributes questionnaire was used to evaluate delayed ratings of participant for individual attributes of FF and MF nasal spray. Number of participants responding to product attributes using delayed attributes questionnaire, Question 9, "Did product cause nasal irritation?" are summarized. The delayed attributes questionnaire was completed 2 minutes after dosing, in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: no; 1: very slightly; 2: slightly; 3: neither slightly nor moderately; 4: moderately; 5; markedly; 6: very markedly. Delayed attribute ratings were analyzed using an analysis of variance mixed model with participant as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of delayed attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Approximatly two minutes after the dosing in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  None | 211 | 172
  Very slight | 45 | 60
  Slight | 16 | 26
  Neither slight nor moderate | 3 | 8
  Moderately | 0 | 6
  Marked | 1 | 4
  Very marked | 0 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Median Difference (Final Values) = 0.00

21. Secondary Outcome: Number of Participants Responding to the Delayed Attributes Question Regarding Bothersome Nasal Irritation.
Description: Delayed attributes questionnaire was used to evaluate delayed ratings of participant for individual attributes of FF and MF nasal spray. Number of participants responding to product attributes using delayed attributes questionnaire, Question 10, "How bothersome was nasal irritation?" are summarized. The delayed attributes questionnaire was completed 2 minutes after dosing, in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: none; 1: very slightly; 2: slightly; 3: neither slightly nor moderately; 4: moderately; 5; markedly; 6: very markedly. Delayed attribute ratings were analyzed using an analysis of variance mixed model with participant as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of delayed attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Approximatly two minutes after the dosing in Period 1 and 2
Population: PP Population. Only participants responded to the question were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 71 | 103
Participants
  None | 19 | 11
  Very slightly | 36 | 51
  Slightly | 14 | 26
  Neither slightly nor moderately | 2 | 5
  Moderately | 0 | 9
  Markedly | 0 | 1
  Very markedly | 0 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Median Difference (Final Values) = 0.00

22. Secondary Outcome: Number of Participants Responding to the Delayed Attributes Question Regarding Satisfaction With Product.
Description: Delayed attributes questionnaire was used to evaluate delayed ratings of participant for individual attributes of FF and MF nasal spray. Number of participants responding to product attributes i.e. taste, using delayed attributes questionnaire, Question 11, "How satisfied with product?" are summarized. The delayed attributes questionnaire was completed 2 minutes after dosing, in Period 1 and 2. Participants specified their responses on a 6-point scale: 0: very satisfied; 1: moderately satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied; 5; moderately dissatisfied; 6: very dissatisfied. Delayed attribute ratings were analyzed using an analysis of variance mixed model with participant as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of delayed attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Approximatly two minutes after the dosing in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  Very satisfied | 104 | 75
  Moderately satisfied | 66 | 83
  Somewhat satisfied | 43 | 52
  Neither satisfied nor dissatisfied | 44 | 45
  Somewhat dissatisfied | 11 | 12
  Moderately dissatisfied | 3 | 6
  Very dissatisfied | 5 | 3
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 0.568, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Median Difference (Final Values) = 0.00

23. Secondary Outcome: Number of Participants Responding to the Delayed Attributes Question Regarding Likeliness to Comply if Prescribed
Description: Delayed attributes questionnaire was used to evaluate delayed ratings of par. for individual attributes of FF and MF nasal spray. Number of par. responding to product attributes i.e. taste, using delayed attributes questionnaire, Question 12, "How likely to comply if prescribed?" are summarized. The delayed attributes questionnaire was completed 2 minutes after dosing, in Period 1 and 2. Par. specified their responses on a 6-point scale: 0: very likely; 1: moderately likely; 2: somewhat likely; 3: neither likely nor unlikely; 4: somewhat unlikely; 5; moderately unlikely; 6: very unlikely. Delayed attribute ratings were analyzed using an analysis of variance mixed model with participant as a random effect, and country, treatment, period, and Baseline rhinitis symptomatology subgroup, and treatment sequence as main effects. P-values associated with tests of delayed attribute rating scores were adjusted for multiplicity using Hochberg's method.
Time Frame: Approximatly two minutes after the dosing in Period 1 and 2
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | MF 200 µg
Number analyzed (Participants) | 276 | 276
Participants
  Very likely | 151 | 128
  Moderately likely | 51 | 67
  Somewhat likely | 37 | 50
  Neither likely nor unlikely | 19 | 13
  Somewhat unlikely | 5 | 11
  Moderately unlikely | 4 | 5
  Very unlikely | 9 | 2
Statistical Analysis 1: Comparison: FF 110 µg vs MF 200 µg; Test type: Superiority or Other; p = 0.951, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Median Difference (Final Values) = 0.00

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of study treatment until the follow-up contact (up to 96 hours).
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who were randomized to treatment.
Arm/Group | FF 110 µg | MF 200 µg
Serious Adverse Events (participants affected / at risk) | 0/298 | 0/298
Other Adverse Events (participants affected / at risk) | 1/298 | 5/298
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF 110 µg (N=298) | MF 200 µg (N=298)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.